Efficacy and safety of moxidectin-albendazole combination for *Trichuris trichiura* infections in school-aged children: a double-blind randomised controlled superiority trial

**NCT Number: NCT06188715** 

Document date: 02 April 2024

Efficacy and safety of moxidectin-albendazole combination for *Trichuris* trichiura infections in school-aged children: a double-blind randomised controlled superiority trial

| <b>Document Version</b> | 1 | <b>Document Date</b> | 02 April 2024 |
|---|---|---|---|
| | Prof. Dr. Jennifer Ke | iser, | |
| | Swiss Tropical and P | ublic Health Institute, | |
| <b>Sponsor Contact</b> | Tel.: +41 61 284 82 1 | 8 | |
| | Fax: +41 61 284 81 0 | 05 | |
| | E-mail: jennifer.keise | er@unibas.ch | |
| | Prof. Dr. Jennifer Ke | iser, | |
| | Swiss Tropical and P | ublic Health Institute, | |
| Principle Investigator | Tel.: +41 61 284 82 1 | 8 | |
| | Fax: +41 61 284 81 0 | 05 | |
| | E-mail: jennifer.keise | er@unibas.ch | |
| <b>Funding Agency</b> | Swiss National Scien | ce Foundation | |

# 1. General information

# I. List of investigators and other persons involved

| Title | Names | Institution | Position | Function in trial |
|---|---|---|---|---|
| Prof. Dr. | Jennifer Keiser | Swiss Tropical and | Unit head | Principal |
| | | Public Health | | Investigator |
| | | Institute (Swiss | | |
| | | TPH), Allschwil, | | |
| | | Switzerland | | |
| MSc | Said Mohammed | Public Health | CEO | Co-PI |
| | Ali | Laboratory Ivo de | | |
| | | Carneri (PHL-IdC) | | |
| | | Foundation, Pemba, | | |
| | | Tanzania | | |
| Dr. | Ibrahim Said | Ministry of Health, | Project leader, | Study physician |
| | Mohammed | Pemba, Tanzania | physician | |
| MSc | Viviane Sprecher | Swiss TPH, | Doctoral student | Co-PI, |
| | | Allschwil, | | Study pharmacist |
| | | Switzerland | | |
| MSc | Annina Schnoz | Swiss TPH, | Doctoral student | Co-PI |
| | | Allschwil, | | |
| | | Switzerland | | |
| Dr. | Jan Hattendorf | Swiss TPH, | Project leader | Statistician |
| | | Allschwil, | | |
| | | Switzerland | | |

# II. Signatures

# **Principal investigator**

| Signature & Date | Docusigned by: Junifor keiser EBEBBS4879400. |
|---|---|
| Name | Jennifer Keiser |
| Title | Prof. Dr. |
| Institution | Swiss Tropical and Public Health Institute |
| Address | Department of Medical Parasitology and Infection Biology |
| | Swiss Tropical and Public Health Institute, Kreuzstrasse 2 |
| | CH-4123 Allschwil, Switzerland |
| Phone | +41 61 284 82 18 |

#### Statistician

| Signature & Date | Docusigned by: 02-Apr-2024 17:26:00 CET A000A7891803407 |
|---|---|
| Name | Jan Hattendorf |
| Title | Dr. |
| Institution | Swiss Tropical and Public Health Institute |
| Address | Department of Epidemiology and Public Health |
| | Swiss Tropical and Public Health Institute, Kreuzstrasse 2, |
| | CH-4123 Allschwil, Switzerland |
| Phone | +41 61 284 81 93 |

I have read this protocol and agree that it contains all necessary details for carrying out this trial. I will conduct the trial as outlined herein and will complete the trial within the time designated.

I will provide copies of the protocol and all pertinent information to all individuals responsible to me who assist in the conduct of this trial. I will discuss this material with them to ensure they are fully informed regarding the drug and the conduct of the trial.

I will use only the informed consent forms approved by the Sponsor or its representative and will fulfil all responsibilities for submitting pertinent information to the Independent Ethics Committees responsible for this trial.

I agree that the Sponsor or its representatives shall have access to any source documents from which Case Report Form information may have been generated.

# **Co-Principal investigator**

| Signature & Date | Sufely |
|------------------|-----------------------------------------|
| Name | Said Mohammed Ali |
| Title | MSc |
| Institution | Public Health Laboratory Ivo de Carneri |
| Address | P.O. Box 122 Wawi, Chake Chake, |
| | Pemba, Tanzania |
| Phone | +255 24 245 20 03 |

# Study physician

| Signature & | 400 |
|-------------|---------------------------------|
| Date | Dung in |
| Name | Ibrahim Said Mohammed |
| Title | Dr. |
| Institution | Ministry of Health Pemba |
| Address | P.O. Box 122 Wawi, Chake Chake, |
| | Pemba, Tanzania |
| Phone | +255 77 253 05 31 |

# Co-Principal investigator, Study pharmacist

| Signature & Date | O2-Apr-2024 17:54:08 CET |
|---|---|
| Name | Viviane Sprecher |
| Title | MSc |
| Institution | Swiss Tropical and Public Health Institute |
| Address | Department of Medical Parasitology and Infection Biology |
| | Swiss Tropical and Public Health Institute, Kreuzstrasse 2 |
| | CH-4123 Allschwil, Switzerland |
| Phone | +41 61 284 92 44 |

# Co-Principal investigator

| Signature & | DocuSigned by: 02-Apr-2024 17:46:44 CET |
|-------------|------------------------------------------------------------|
| Date | lnuina Souron 02-Apr-2024 17:48:44 CET |
| Name | Annina Schnoz |
| Title | MSc |
| Institution | Swiss Tropical and Public Health Institute |
| Address | Department of Medical Parasitology and Infection Biology |
| | Swiss Tropical and Public Health Institute, Kreuzstrasse 2 |
| | CH-4123 Allschwil, Switzerland |
| Phone | +41 61 284 92 86 |

# **Table of contents**

| 1. | Gen | eral information | 2 |
|----|-------|------------------------------------------------|----|
| 2. | Bacl | kground information | 13 |
| 3. | Tria | l objective and purpose | 14 |
| 4. | Met | hodology | 15 |
| | 4.1 | Primary and secondary endpoint | 15 |
| | 4.2 | Trial design | 15 |
| | 4.3 | Procedures | 16 |
| | 4.3. | 1 Diagnosis | 16 |
| | 4.3.2 | 2 FECPAKG2 | 16 |
| | 4.3.3 | 3 Clinical examination | 17 |
| | 4.3.4 | 4 Treatment of participants | 17 |
| | 4.3.5 | 5 Pharmacokinetic analysis | 18 |
| | 4.3.0 | Safety assessment | 19 |
| | 4.3.7 | 7 Efficacy assessment | 19 |
| | 4.4 | Measure to minimise bias | 19 |
| | 4.5 | Study duration and duration of participation | 19 |
| 5. | Sele | ction of trial participants | 20 |
| | 5.1 | Recruitment | 20 |
| | 5.2 | Inclusion criteria. | 20 |
| | 5.3 | Exclusion criteria | 21 |
| | 5.4 | Criteria for discontinuation of trial. | 21 |
| | 5.5 | Concomitant medication | 21 |
| 6. | Safe | ety assessments | 21 |
| | 6.1 | Adverse event definitions | 22 |
| | 6.1. | 1 Severity grading | 22 |
| | 6.1.2 | 2 Relatedness | 23 |
| | 6.1.3 | 3 Expectedness | 23 |
| | 6.1.4 | 4 Serious adverse events | 23 |
| | 6.1.5 | Suspected unexpected serious adverse reactions | 24 |

| 6.2 | Methods of recording and assessing adverse events | 24 |
|---|---|---|
| 6.3 | Reporting of serious adverse events | 25 |
| 6.4 | Safety reporting to Health Authorities, Ethics Committees and other third parties | 25 |
| 6.5 | Rescue medication strategy | 26 |
| 7. I | Data management and data quality control | 26 |
| 7.1 | Source data | 26 |
| 7.2 | Data collection and documentation | 26 |
| 7.3 | Ethical, legal and security issues | 27 |
| 7.4 | Data storage and preservation | 27 |
| 7.5 | Study documents: translations – reference language | 28 |
| 8. S | Statistics | 28 |
| 8.1 | Definition of primary endpoint | 28 |
| 8.2 | Justification of number of trial participants | 28 |
| 8.3 | Description of statistical methods | 28 |
| 9. I | Outies of the investigator | 30 |
| 9.1 | Investigator's confirmation | 30 |
| 9.2 | Damage coverage | 30 |
| 9.3 | Project management | 30 |
| 10. | Ethical considerations | 31 |
| 10. | 1 Independent Ethics Committee (IEC) | 31 |
| 10.2 | 2 Evaluation of the risk-benefit ratio | 31 |
| 10 | Participant information and consent | 31 |
| 10.4 | 4 Participants requiring particular protection | 32 |
| 11. | Quality control and quality assurance | 32 |
| 11. | 1 Monitoring and auditing | 32 |
| 11.2 | Data and safety monitoring board (WHO) / data monitoring committee (EU/FDA) | 32 |
| 12. | Funding. | 33 |
| 13. | Dissemination of results and publication | 33 |
| 14 | References | 34 |

III. Abbreviations

AE Adverse event

CI Confidence interval

CR Cure rate

CRF Case report form

EKNZ Ethikkommission Nordwest- und Zentralschweiz

EPG Eggs per gram

ERR Egg reduction rate

EU European Union

FDA Food & Drug Administration

GCP Good clinical practice

Hb Haemoglobin

ICF Informed consent form

ICH International council for harmonization of technical requirements for

pharmaceuticals for human use

IEC Independent ethics committee

MDA Mass drug administration

NLME nonlinear mixed-effects

PC Preventive chemotherapy

PHL-IdC Public Health Laboratory Ivo de Carneri

PI Principal investigator

PK Pharmacokinetics

SAC School-aged children

SAE Serious adverse event

SNSF Swiss National Science Foundation

STH Soil-transmitted helminths

SUSAR Suspected unexpected serious adverse reaction

Swiss TPH Swiss Tropical and Public Health Institute

WHO World Health Organization

# IV. Synopsis

| Sponsor/Sponsor- | Prof. Dr. Jennifer Keiser |
|---|---|
| Investigator | |
| Study title | Efficacy and safety of moxidectin-albendazole combination for <i>Trichuris trichiura</i> infections in school-aged children: a double-blind randomised controlled superiority trial |
| Short title | Moxidectin-albendazole combination for <i>Trichuris trichiura</i> —infected children |
| Study acronym | Moxiped |
| Protocol version and date | v1, 02 April 2024 |
| Trial registration | Registered on <a href="https://www.clinicaltrials.gov/">https://www.clinicaltrials.gov/</a> (NCT06188715) |
| Clinical phase | Phase 3 trial |
| Sample size | 210 participants |
| Indication | Trichuris trichiura infection (eggs in stool) |
| Investigational and reference treatment | Moxidectin-albendazole combination Reference: albendazole and placebo |
| Study rationale | To provide evidence on the efficacy and safety of co-administered moxidectin and albendazole compared to albendazole monotherapy in school-aged children (SAC; aged 6-12 years) infected with <i>T. trichiura</i> . Additionally, to substantiate evidence on the safety profile of moxidectin-albendazole combination in this age group using a placebo (and albendazole) only arm. To date, this has only been established in adolescents (aged 16-18 years), who might present different symptoms or symptom severity compared with SAC. |

| Study objectives | Our <b>primary objective</b> is to demonstrate superiority of |
|---|---|
| | a) Arm A: moxidectin (4 mg / 8 mg) & albendazole (400 mg) |
| | combination, |
| | compared to |
| | b) Arm B: albendazole (400 mg) |
| | in terms of cure rate (CR), assessed at 14-21 days post-treatment by |
| | quadruplicate Kato-Katz microscopy, in SAC (6-12 years) infected with |
| | T. trichiura. |
| | The <b>secondary objectives</b> of the trial are: |
| | a) to determine the <i>T. trichiura</i> egg reduction rates (ERRs) of treatments; |
| | b) to determine the CRs and ERRs of treatments against |
| | Ascaris lumbricoides and hookworm co-infection; |
| | c) to evaluate the safety and tolerability of the treatments; |
| | d) to characterize population pharmacokinetics (PK) of moxidectin |
| | in <i>T. trichiura</i> infected SAC. |
| | The <b>exploratory objective</b> of this trial is to assess the diagnostic |
| | performance of FECPAKG2. |
| Study design | Parallel randomised controlled superiority trial |
| Study product / | Administration of a single oral dose of moxidectin (4 mg or 8 mg) and |
| intervention | albendazole (400 mg) |
| Comparator(s) | Albendazole (400 mg), placebo |
| Key inclusion / Exclusion | Inclusion: |
| criteria | • Individuals aged 6-12 years (confirmed by birth certificate or |
| | similar document); |
| | • having given written informed consent signed by |
| | parents/caregivers and assent by participant; |
| | being able and willing to provide two stool samples at baseline |
| | and at follow-up assessment (14-21 days); |
| | • having at least two out of four Kato-Katz slides positive for |
| | T. trichiura at baseline; |
| | • being able and willing to be examined by a study physician |
| | before and after treatment. |

| | Exclusion: |
|---|---|
| | <ul> <li>presence or signs of major systemic illness, e.g. fever (temporal body temperature of &gt;38.0°C), severe anaemia (haemoglobin level of &lt;80 g/l);</li> <li>history of severe acute disease or unmanaged, severe chronic disease (i.e., condition is not as therapeutically controlled as necessary);</li> <li>use of anthelminthic drugs during study period;</li> <li>known allergy to study medication (i.e., moxidectin or albendazole);</li> <li>being prescribed or taking concomitantly medication with known contraindications or drug interactions with the study medication;</li> <li>pregnancy (female participants aged 10-12 years);</li> <li>concurrent participation in other clinical trials.</li> </ul> |
| Primary endpoints | • <i>T. trichiura</i> infection status of participants at 14-21 days post-treatment assessed by quadruplicate Kato-Katz |
| Secondary endpoints | <ul> <li>T. trichiura infection intensity of participants at 14-21 days post-treatment assessed by quadruplicate Kato-Katz</li> <li>A. lumbricoides and hookworm infection status and intensity of co-infected participants at 14-21 days post-treatment assessed by quadruplicate Kato-Katz</li> <li>Adverse events (AEs)</li> <li>Population PK parameters of moxidectin in T. trichiura infected SAC</li> </ul> |
| Exploratory endpoints | Diagnostic characteristics of FECPAKG2 (infection intensity, sensitivity, and specificity) compared to Kato-Katz |
| Interim analyses | None |
| Study duration | 2 months |
| Schedule | 04/2024: of first participant in (planned) 06/2024: of last participant out (planned) |

| Study centres | T. trichiura endemic villages, Wete district, Pemba Island, Tanzania |
|---|---|
| Measurements & | For the initial diagnosis and efficacy assessment at 14-21 days post- |
| procedures | treatment, two stool samples will be collected from each participant on |
| | two consecutive days. All stool samples will be examined for presence |
| | of T. trichiura, A. lumbricoides, and hookworm eggs with duplicate |
| | Kato-Katz thick smears assessed via bright-field microscopy. The |
| | medical history of the participants will be assessed with a standardised |
| | questionnaire, in addition to a clinical examination carried out by the |
| | study physician before treatment. All participants will be interviewed |
| | before treatment and at three and 24 hours and 14-21 days post-treatment |
| | for the occurrence of AEs. Any potential AEs happening between 3 |
| | hours and the respective follow-up time points will be monitored by |
| | local healthcare workers and medical intervention provided if necessary. |
| | Each participant will be asked to provide a finger-prick blood sample for |
| | haemoglobin measurement at baseline. At the same time, |
| | anthropometric measurements (i.e. height, and weight) will be taken for |
| | all participants. In addition, female participants aged 10-12 years will be |
| | asked to provide a urine sample to determine pregnancy. |
| | To determine PK parameters of moxidectin, a subsample of 12 study |
| | participants per moxidectin dose (4 mg and 8 mg) will be asked to |
| | provide a maximum of 5 micro blood samples per participant using |
| | finger pricks at defined time points between 1 hour and 24 hours. |
| Statistical analyses | An available case analysis (full analysis set according to the intention to |
| | treat principles) will be performed, including all participants with |
| | primary endpoint data. Additionally, a per-protocol analysis will be |
| | conducted. CRs will be calculated as the percentage of egg-positive |
| | participants at baseline who become egg-negative after treatment. |
| | Differences in CRs (between treatment arms) will be analysed using |
| | logistic regression. |
| | Geometric and arithmetic mean egg counts will be calculated for the |
| | different treatment arms before and after treatment to assess the |
| | corresponding ERRs. Bootstrap resampling with 5,000 replicates will be |
| | used to calculate 95% confidence intervals (CIs) for ERRs and |

| | AEs will be compiled into frequency tables and compared between |
|---|---|
| | treatment groups using descriptive summary statistics. |
| | With regard to population PK parameters, Cmax and tmax will be |
| | observed values, AUC and $t_{1/2}$ will be calculated using nonlinear mixed- |
| | effects (NLME) modelling with the WinNonlin software package. In |
| | addition, exploratory pharmacometric PK and exposure-response |
| | analyses may be performed with the Monolix or NONMEM software |
| | package. |
| GCP statement | This study will be conducted in compliance with the protocol, the current |
| | version of the Declaration of Helsinki, ICH-GCP E6 (R2) as well as all |
| | national legal and regulatory requirements. |
| Key explanation for the | This study will involve children aged 6-12 years, since an infection with |
| inclusion of children | T. trichiura occurs most often in children who are therefore the main |
| | target group of deworming campaigns. The main goal of the study is to |
| | evaluate for the first time the efficacy and safety of moxidectin- |
| | albendazole in this age group. |
| Recruitment procedure | The trial will be conducted on Pemba Island, Tanzania. It will take place |
| | in areas with moderate to high <i>T. trichiura</i> endemicity (communities |
| | with a prevalence of ≥20%) identified from earlier studies and/or based |
| | on experience of the local collaborating team. |
| Coverage of damages | Winterthur Insurance, Policy No. 4746321; |
| | Pemba: National Insurance Cooperation of Tanzania LTD, Policy No. |
| | IMIS/GL/P/25/1/2024/771417 |
| Storage of data and | After the study has been completed, all samples will be destroyed. Case |
| samples for future | report forms and electronic source data will be kept for a minimum of |
| research aims | 15 years. |
| ~ ~ | |
| Conflict of interest in | We declare no conflict of interest in relation to the investigated drugs. |
| relation to the investigated | |
| drugs | |

# 2. Background information

Trichuriasis is a parasitic disease caused by nematodes belonging to the group of soil-transmitted helminths (STH). It is estimated that around 400 million people harbour infections with *Trichuris trichiura* globally [1]. As it is the case for all STH infections, trichuriasis is mainly endemic in developing countries in tropical and subtropical regions, with highest burden among rural communities due to its link to poor sanitation [2].

Infection with *T. trichiura* occurs when ingesting embryonated eggs via soil-contaminated hands, drinking water or food. Having reached the small intestine, the eggs hatch realising the larvae. The larvae migrate directly into the cecum where they develop into adult worms and begin to oviposit. Eggs are excreted into the soil via the faeces, thereby closing the life cycle [3].

Acute symptoms of trichuriasis are generally mild or not apparent in infected individuals living in endemic areas [2, 4]. The main disease burden results from chronic infection and repeated re-infection, in which symptoms related to the location of adult worms such as abdominal pain may develop. Long-term infection compromises the life of people by hampering their physical and mental development, limiting their work performance and overall quality of life [4].

The recent World Health Organization (WHO) road map for neglected tropical diseases targets STH infections for near to global elimination as a public health problem by 2030 [5]. One important intervention to achieve this is preventive chemotherapy (PC) [5-7]. The aim of PC is to reduce worm burden and hence morbidity in endemic populations by regular large-scale administration of anthelminthic drugs to high-risk groups, *e.g.* preschool-aged and school-aged children (SAC) [8, 9]. The frequency of such mass drug administration (MDA) depends on the local infection prevalence [8, 9]. At present, the benzimidazoles albendazole and mebendazole are the most widely used drugs for PC campaigns against STH infections [7, 10]. These drugs are characterized by high cure rates (CRs) against infections with *Ascaris lumbricoides* (>95%) and moderate CRs against hookworm infections (80%). However, at single oral doses suitable for MDA, these drugs have demonstrated unsatisfactory efficacy against *T. trichiura* infections [11, 12].

Therapies combining two or more drugs are widely advocated in different therapeutic areas. The advantages of multifactorial pharmacological treatment include the increase and broadening of efficacy over drugs being administered in monotherapy and the protection against the selection of drug resistance, and hence, a prolongation of the life-span of effective and available drugs [13-15]. In 2017, ivermectin in combination with albendazole for treatment of STH was added to the Essential Medicines List (EML) paving the way to further evaluate the efficacy of combination treatments among SAC and communities in a range of epidemiological settings [16].

Moxidectin, a macrocyclic lactone like ivermectin, has been approved by the United States Food & Drug Administration (FDA) for the treatment of onchocerciasis in 2018 in individuals aged  $\geq$ 12 years [17]. The combination of moxidectin (at a dose of 8 mg) and albendazole has shown promising efficacy

against T. trichiura infections in adolescents and adults [18-20]. However, there is a need to explore whether moxidectin could reveal a benefit in the treatment of STH infections in SAC. A phase 1 trial determining safety and pharmacokinetics of moxidectin in children aged 4-11 years living in Ghana has recently been completed [21]. Based on the findings of this trial, it was recommended to administer single doses of 4 mg moxidectin to individuals aged  $\leq$ 8 years and 8 mg to individuals aged  $\geq$ 8 years. In this trial, we aim to evaluate if the recommended doses of moxidectin in combination with albendazole are a safe and efficacious treatment against T. trichiura infection in SAC on Pemba Island, Tanzania, and superior to albendazole monotherapy. Furthermore, given that the most commonly reported adverse events of moxidectin and albendazole correspond to the main symptoms of trichuriasis, a placebo only arm will be included to better define the safety profile of moxidectin-albendazole combination. To date, this has only been established in adolescents (aged 16-18 years), who might present different symptoms or symptom severity compared with SAC.[18] Finally, we re-assess pharmacokinetic (PK) parameters of moxidectin in SAC. The PK characterization of a drug is essential to understand the response of the human body to a drug and vice versa, especially in populations that physiologically differ from healthy adults. Physiological characteristics like mal- or undernutrition due to intestinal worms, such as T. trichiura, can potentially affect the PK of a drug [22, 23]. Age, sex, bodyweight but also the presence of certain enzymes in different populations are important contributors to the PK profile of a drug. Our study will be the first one to provide PK information on moxidectin in SAC with trichuriasis and thus guide optimal drug dosing in this high-risk population.

# 3. Trial objective and purpose

We designed a superiority trial to show that moxidectin-albendazole combination is superior compared to albendazole monotherapy in treating trichuriasis in individuals aged 6-12 years on Pemba Island, Tanzania. This study will provide further insights on the value of moxidectin-albendazole combination. Our data will support the development of moxidectin in children aged <12 years and its implementation in control programs. As recommended for new combination therapies, we assess superiority of the drug combination compared to standard-of-care monotherapy. In addition, we aim to substantiate evidence on the safety profile of moxidectin-albendazole combination in SAC using a placebo only arm.

The **primary objective** is to demonstrate that co-administered moxidectin (4 mg / 8 mg) & albendazole (400 mg) is superior to albendazole (400 mg) monotherapy in terms of CR in *T. trichiura*-infected children aged 6-12 years assessed at 14-21 days post-treatment by quadruplicate Kato-Katz microscopy.

The **secondary objectives** of the trial are:

- a) to determine the *T. trichiura* egg reduction rates (ERRs) of treatments;
- b) to determine the CRs and ERRs of treatments against *A. lumbricoides* and hookworm co-infection;
- c) to evaluate the safety and tolerability of the treatments;

d) to characterize population PK of moxidectin in T. trichiura infected SAC.

The **exploratory objective** of this trial is to assess the diagnostic performance of FECPAKG2.

# 4. Methodology

## 4.1 Primary and secondary endpoint

**Primary endpoint:** *T. trichiura* infection status of participants at 14-21 days post-treatment assessed by quadruplicate Kato-Katz.

# **Secondary endpoints:**

- *T. trichiura* infection intensity of participants at 14-21 days post-treatment assessed by quadruplicate Kato-Katz;
- *A. lumbricoides* and hookworm infection status and intensity of co-infected participants at 14-21 days post-treatment assessed by quadruplicate Kato-Katz;
- Tolerability of treatments (adverse events (AEs)) at three and 24 hours and 14-21 days post-treatment;
- Population PK parameters of moxidectin in *T trichiura* infected SAC.

**Exploratory endpoints:** Diagnostic characteristics of FECPAKG2 (infection intensity, sensitivity, and specificity) compared to Kato-Katz.

# 4.2 Trial design

A parallel randomised controlled superiority trial will be conducted with three treatment arms (Figure 1). The study includes a baseline screening (day -30 to -1) and clinical baseline assessment (day 0) before treatment and post-treatment assessments for safety (day 0, 1 and 14 to 21) and efficacy (day 14 to 21). It is designed as a parallel three-arm trial with 210 participants aged 6-12 years randomised to either moxidectin (4 mg for 6-7 year-olds and 8 mg for 8-12 year-olds) and albendazole (400 mg), moxidectin placebo and albendazole (400 mg), or moxidectin placebo and albendazole placebo, with an allocation ratio of 3:2:1 (*i.e.*, 105:70:35). This trial will be conducted in communities in the Wete district on Pemba Island with high endemicity as identified in previous studies on *T. trichiura*.



Figure 1. Trial design and timeline.

### 4.3 Procedures

#### 4.3.1 Diagnosis

At baseline, all participants will be asked to provide two stool samples. From each stool specimen, duplicate Kato-Katz thick smears (41.7 mg each) [24] will be prepared and read under a microscope for eggs of *T. trichiura*, *A. lumbricoides* and hookworm by experienced technicians. Eggs per gram (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. For quality control of *T. trichiura* and *A. lumbricoides* egg counts, 10% of slides will be re-read by another laboratory technician. Results are considered correct if the following tolerance margin is not exceeded: (i) No difference in presence/absence of *T. trichiura* and *A. lumbricoides* (ii) egg counts are +/-10 eggs for counts ≤100 eggs or +/-20% for counts >100 eggs (for each species separately). In case discrepancies above the tolerance margin are noted in one or more slides, the respective slides are re-read by the local technicians. The new results are discussed, so that in case of discordant results, slides can be re-evaluated to reach consensus. All microscopically analysed quadruplicate Kato-Katz thick smears will be destroyed after passing the quality control. The same diagnostic approach will be applied at 14-21 days after treatment (see section 4.3.7).

#### 4.3.2 FECPAKG2

Research on new diagnostic tools is necessary, since the currently recommended Kato-Katz technique has a low sensitivity for low STH infections and slides with hookworm eggs cannot be re-examined [25-27]. Once moving towards transmission control and STH elimination, an increased sensitivity of the diagnostic method of choice is crucial [28]. Preferably, a diagnostic method that could potentially

replace Kato-Katz would be sensitive, specific, fast, simple, cost-effective and re-analysis could be conducted at any time.

The aim of this exploratory objective within this trial is the comparison of infection intensity, sensitivity, and specificity of the Kato-Katz technique with the novel diagnostic tool FECPAKG2 (Techion). FECPAKG2 is an online, remote location, parasite diagnostic system used in veterinary medicine [29]. An image of the Kato-Katz slide is captured, stored offline on a computer, and can be uploaded onto a cloud once connected to the internet. Subsequently, specialists around the world can analyse the image at any time. Techion's image capture devices are robust, reliable, versatile and cost effective [30]. Baseline quadruplicate Kato-Katz thick smears will be used to take images by FECPAKG2 after the slides have been read by technicians under the microscope.

#### 4.3.3 Clinical examination

A clinical examination of the study participants assessing general health, anthropometric parameters including height and weight as well as temperature using a non-contact infrared forehead thermometer (Braun No touch – NTF3000; Braun, Kronberg, Germany) will precede the treatment. Each participant will be asked to provide a finger-prick blood sample to measure haemoglobin (Hb) levels, which will be detected using a HemoCue analyzer (Hb 301 system, Angelholm, Sweden). In case of abnormal values, results from baseline clinical examination may be reported back to participants and their parents/caregivers during the trial period. To avoid accidental treatment of pregnant girls, all female participants aged 10-12 years will be asked to provide a urine sample to be subjected to a pregnancy RDT during clinical examination All trial participants will further be asked about existing clinical symptoms before drug administration using a standardised questionnaire.

### 4.3.4 Treatment of participants

All eligible participants will be treated with the respective treatment regimen according to their treatment arm assigned by randomisation at day 0. Moxidectin tablets (2 mg) and appearance-matching placebo tablets will be obtained from Medicines Development for Global Health (MDGH), Australia, and two or four tablets of 2 mg will be administered, depending on the age of participants (two tablets of 2 mg for 6-7 year-olds and four tablets of 2 mg for 8-12 year-olds). Albendazole will be the product of GSK (Zentel®) and a single tablet of 400 mg will be administered. Albendazole placebo tablets will be purchased from Fagron, Germany.

The tablets will be handed out from four drug containers (moxidectin, moxidectin placebo, albendazole and albendazole placebo). According to the randomisation list, each person will receive either:

- (i) Two or four tablets of moxidectin plus a single tablet of albendazole
- (ii) Two or four tablets of moxidectin placebo plus a single tablet of albendazole
- (iii) Two or four tablets of moxidectin placebo plus a single tablet of albendazole placebo

All drugs will be administered in the presence of the Principal Investigator (PI) and/or Co-PI, and ingestion confirmed. This will be recorded with the time and date of dosing. Participants will be asked to limit the use of any drugs other than those prescribed by the study medical team for the duration of the study as described in section 5.5. After ingestion of the medication, the participants will be observed for three hours to ensure retention of the drug. Vomiting within one hour post-dosing will require redosing. The participants will not be allowed more than one repeated dose. No re-administration will be needed for participants vomiting after one hour. The PI or the Co-PIs are responsible for drug accountability at the study site. Maintaining drug accountability includes careful and systematic study drug storage, handling, dispensing, and documentation of administration. Prior to administration, drugs will be stored at room temperature and protected from light and exposure to moisture in a secure area with limited access at the study site.

To avoid interference of potential on-going control programs against helminthiases with the infection status of the trial participants, communication with local stakeholders will be established to ascertain that trial participants will not undergo MDA treatment. Missed-out rounds of planned MDA against STH infections will be substituted with a free single-dose treatment (albendazole 400 mg) against STH infection after the follow-up assessment, offered by the study team to all community members not participating in the trial in communities screened.

#### 4.3.5 Pharmacokinetic analysis

The PK and exposure-response correlation study will be performed in 24 participants in the moxidectinalbendazole arm (12 per moxidectin dose), randomly selected by location. Since PK population parameters of moxidectin are available, a sparse sampling approach can be applied to describe the PK profile [21, 31]. Within a sparse sampling approach, instead of describing the PK profile for each participant separately, samples are allocated to different time points and/or individuals within the same treatment. Statistical inferences are performed to characterize the population-based PK profile of a specific dose. This approach allows for a reduced number of samplings per dose and renders a PK characterization well tolerable. To this end, a small drop of blood from the fingertip will be taken for a maximum of 5 finger pricks per participant. The exact time points are 1h, 2h, 4h, 6h, and 24h, covering the relevant time span identified previously [21, 31]. Capillary blood (~10 µl) will be collected by puncture with a finger prick. Two micro-samples (duplicates) will be taken with one finger prick. Each time, the drop of blood (10 µl) will be directly transferred on Mitra® sticks [31]. The dried sticks will be transported to Swiss TPH and stored at room temperature until analysis (< 2 months post-treatment). The quantification of the study drugs will be performed using the validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method as described elsewhere [31]. Drug concentrations will be calculated by interpolation from a calibration curve with a lower limit of quantification of 1-5 ng/ml. 7% of the sample duplicates will be analysed for quality control, and the measured concentrations will be used to determine between-run and overall precision and accuracy of the analysis.

#### 4.3.6 Safety assessment

Participants will be monitored at the site (*i.e.* school) for three hours after treatment administration to observe any possible acute AEs (continuous observation) and reassessment will be done at 24 hours post-treatment (follow-up visit). Additionally, interviews will be conducted to determine the emergence of clinical symptoms such as headache, abdominal pain, itching, nausea, vomiting and diarrhoea directly before treatment within the scope of baseline assessment. At three and 24 hours and 14-21 days after treatment participants will again be interviewed for the assessment of AEs. Symptoms arising within three hours after treatment and the follow-up time points will be monitored by parents/caregivers, teachers or local healthcare workers who will report incidences to the study team. Any symptoms will be recorded in the designated case report form (CRF) and immediate action will be undertaken if indicated.

## 4.3.7 Efficacy assessment

The efficacy of the treatment will be determined at 14-21 days post-treatment by collecting another two stool samples, which will be microscopically examined for *T. trichiura*, *A. lumbricoides* and hookworm eggs using quadruplicate Kato-Katz thick smears (two slides per sample). Quality control will be performed as described for the initial diagnosis (see section 4.3.1). All microscopically analysed quadruplicate Kato-Katz thick smears will be destroyed after passing the quality control.

Participants will be considered cured for an infection if no corresponding eggs are found in the followup stool samples. At the end of the study, all participants remaining positive for *T. trichiura* or any coinfection will be treated with the currently best recommended treatment.

#### 4.4 Measure to minimise bias

Study participants eligible for treatment will be randomly assigned to one of the three treatment arms using a computer-generated stratified randomisation code. The random allocation sequence with random block sizes of 6 and 12 and stratified by two levels of age category (6-7 years and 8-12 years) and two levels of baseline *T. trichiura* infection intensity (light: 1-999 EPG, and moderate or heavy: ≥1000 EPG) will be provided by a statistician. Allocation concealment will be warranted using opaque, sealed envelopes containing the randomisation lists. All treatment arms will be double-blinded (*i.e.* study participants and trial team members assessing the outcomes will be blinded) using appearance-matching placebos. In the case of accidental unblinding or necessary code breaks, the sponsor will be immediately notified (within 24 hours) and data will be analysed as set forth in section 8.3.

### 4.5 Study duration and duration of participation

The trial will last two months. Baseline screening is scheduled to start one month prior to treatment and follow-up stool sample collection will take place at 14-21 days after treatment, lasting approximately two weeks. Thus, the maximum time for participation will be two months. Schedules of visits are summarised in Table 1.

**Table 1.** Schedule of study visits.

| | Screening | Baseline/Treatment/Safety | | | | | Follow up | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Day -30 to -1 | | Day 0 | | | | | Day 14 to 21 | | |
| | | 0h | 42 | 1h | 2h | 3h | 4h | 6h | 24h | |
| Informed consent | X | | and treatment | | | | | | | |
| Diagnosis (stool examination) | X | | trea | | | | | | | X |
| Medical history | | X | | | | | | | | |
| Clinical examination | | X | atior | | | | | | | |
| Haemoglobin measurement | | X | lomis | | | | | | | |
| PK (microsampling) | | | Randomisation | X | X | | X | X | X | |
| Capturing AEs and SAEs | | | | | | X | | | X | X |

# 5. Selection of trial participants

### 5.1 Recruitment

The trial will be carried out in children aged 6-12 years in the Wete district, Pemba Island, Tanzania. The trial will be implemented as school-based study in communities with endemicity of *T. trichiura* infection above 20% identified during previous trials. Parents/caregivers of potential participants will be invited to participate in an information session. The research team will explain the purpose and procedures of the study, as well as potential benefits and risks of participation. Attendees will be encouraged to ask questions which will be discussed in an open setting.

Parents/caregivers interested in having their child participate in the study will be invited to complete the informed consenting process by signing the informed consent form (ICF). In addition, participants will be asked to sign an assent form. Participants having a signed ICF and assent form will be assessed for eligibility during screening procedures.

#### 5.2 Inclusion criteria

- 1. Aged between 6 and 12 years (confirmed by birth certificate or similar document).
- 2. Written informed consent signed by parents/caregivers and assent by participant.
- 3. Agree to comply with study procedures, including provision of two stool samples at the beginning (baseline) and at follow-up assessment 14-21 days after treatment.
- 4. At least two slides of the quadruplicate Kato-Katz thick smears positive for *T. trichiura*.
- 5. Willing to be examined by a study physician prior to treatment.

#### 5.3 Exclusion criteria

- 1. Presence or signs of major systemic illness, e.g. fever (temporal body temperature  $\geq 38^{\circ}$ C) or severe anaemia (Hb level <80 g/l according to WHO [32]) upon initial clinical assessment.
- 2. History of severe acute disease or unmanaged, severe chronic disease (*i.e.*, condition is not as therapeutically controlled as necessary).
- 3. Use of anthelminthic drugs during study period.
- 4. Known allergy to study medication (*i.e.* moxidectin, albendazole).
- 5. Being prescribed or taking concomitantly medication with known contraindication or drug interactions with the study medication.
- 6. Pregnancy (female participants aged 10-12 years).
- 7. Concurrent participation in other clinical trials.

#### 5.4 Criteria for discontinuation of trial

A participant can be discontinued from the study for the following reasons:

- 1. Withdrawal from the study (this can happen anytime as participation is voluntary and there are no further obligations once a participant withdraws).
- 2. At the discretion of the PI or Co-PI, if the participant is not compliant to the requirements of the protocol.

Discontinued participants will not be replaced. If, for any reason, a participant is discontinued from the study before the end of treatment evaluations, the AE assessment will still be conducted. Data obtained prior to the withdrawal will be included in the analysis to ensure the validity of the trial. Data of withdrawn participants are fully anonymised once analysis is complete.

#### 5.5 Concomitant medication

All medications taken between one month before treatment and the follow-up assessment at 14-21 days post-treatment must be recorded with indication, dose regimen, date and time of administration.

Medication(s)/treatment(s) permitted during the trial:

- Analgesics and antipyretics are allowed to be given to participants in case of fever, antiemetics to prevent nausea and vomiting and/or antibiotics to prevent or treat bacterial superinfection.

Medication(s)/treatment(s) NOT permitted during the trial:

- No other active drugs against helminths are permitted during the trial. Participants receiving active anthelminthic concomitant medication during the trial will not be discontinued; however, a case-specific assessment will be done at the point of data analysis.

# 6. Safety assessments

#### 6.1 Adverse event definitions

The term "adverse event" (AE) is defined as follows:

Any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.

An AE could therefore include any of the following events, which develop or increase in severity during the course of the study, after administration of the study product:

- a. Any unfavourable and unintended signs, symptoms or disease temporally associated with the use of a medicinal product, whether or not considered related to the condition under study and the study product.
- b. Any abnormality detected during physical examination.

The medical conditions present at the initial trial visit that do not worsen in severity or frequency during the trial will not be defined as AEs, but considered as baseline medical conditions. For the purpose of this trial, disease progression and relapse will be considered as failure of prescribed treatment or failure of treatment administration, not as an AE.

The observation time for AEs starts when the treatment is initiated until the end of the study.

These data will be recorded on the appropriate CRF sections, regardless of whether they are thought to be associated with the study or the drug under investigation. Associated with the use of the drug means that there is a reasonable possibility that the event may have been caused by the drug (see also relatedness definitions below).

#### 6.1.1 Severity grading

Adverse signs or symptoms will be graded by the physician or nurse of the trial as mild, moderate, severe or life threatening according to the following definitions:

| Grade | Definition |
|---|---|
| 1 | Mild: the participant is aware of the event or symptom, but the event or symptom is easily tolerated. |
| 2 | <u>Moderate</u> : the participant experiences sufficient discomfort to interfere with or reduce his or her usual level of activity. |
| 3 | <u>Severe</u> : significant impairment of functioning: the participant is unable to carry out his or her usual activities. |
| 4 | Life-threatening or disabling |
| 5 | Death related to AEs |

#### 6.1.2 Relatedness

Relatedness will be assessed as defined below based on the temporal relationship between the AE and the treatment, known side effects of treatment, medical history, concomitant medication, course of the underlying disease and trial procedures.

<u>Possibly related</u>: an AE, which can medically (pharmacologically/clinically) be attributed to the study treatment.

<u>Unrelated</u>: an AE, which is not reasonably related to the study treatment. A reasonable alternative explanation must be available.

An AE that is determined to be related to the administration of a study product is referred to as an "adverse drug reaction".

### 6.1.3 Expectedness

<u>Expected adverse drug reaction:</u> Any AE possibly related to the administration of moxidectin, albendazole or moxidectin-albendazole combination reported in the literature or on the drug package leaflets, if available, and listed in the consent form.

<u>Unexpected adverse drug reaction:</u> Any AE possibly related to the study drug administration, the nature, frequency, specificity or severity of which is unanticipated and not consistent with the available risk information described for these drugs.

#### 6.1.4 Serious adverse events

According to the ICH "Clinical Safety Data Management: Definitions and standards for expedited Reporting E2A" [33], a serious adverse event (SAE) includes any event (experience) or reaction in any untoward medical occurrence that at any dose:

- 1. results in death;
- 2. is life-threatening, meaning, the participant was, in the view of the Investigator, at immediate risk of death from the reaction as it occurred, *i.e.* it does not include a reaction that, had it occurred in a more serious form, might have caused death;
- 3. results in persistent or significant disability/incapacity, *i.e.* the event causes a substantial disruption of a person's ability to conduct normal life functions;
- 4. requires inpatient hospitalization or prolongation of existing hospitalization;
- 5. creates a congenital anomaly or birth defect (not relevant for this study);
- 6. is an important medical event, based upon appropriate medical judgement, that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes defining serious.

A "severe" AE does not necessarily meet the criteria for a "serious" AE. SAEs are reported from treatment until the end of the study.

SAEs that are still ongoing at the end of the study period will be followed up to determine the final outcome.

The causality of any SAE that occurs after the study period and its possible relatedness to the study treatment or study participation will also be assessed by investigators as described in section 6.1.2.

# 6.1.5 Suspected unexpected serious adverse reactions

A suspected unexpected serious adverse reaction (SUSAR) is an unexpected adverse drug reaction, which also meets the definition of SAE.

## 6.2 Methods of recording and assessing adverse events

Few AEs have been reported following moxidectin, albendazole, or moxidectin-albendazole co-administration in STH infected individuals. The most common AEs were abdominal cramps, headache, fatigue, nausea, diarrhoea, fever, and vertigo. Such symptoms can, however, also result from the infection itself. Such side effects may be more frequent and/or serious in patients with a heavy worm burden.

The observation time for AEs starts when the treatment is initiated. Participants will be observed for at least three hours following treatment for any acute AE and reassessment will be done at 24 hours and 14-21 days post-treatment. If there is any abnormal finding, the local study physician will perform a full clinical examination and findings will be recorded. An emergency kit will be available on site to treat any medical conditions that warrant urgent medical intervention. Participants will also be interviewed at three and 24 hours as well as at 14-21 days after treatment about the occurrence of AEs. Any potential AEs happening between three hours post-treatment and the further follow-up time points (24 hours and 14-21 days) will be monitored and managed with the help of the locally based medical team (including specifically trained community health workers, nurses and medical doctors). Medical intervention will be provided if necessary.

Information on all AEs (incidence, intensity, seriousness and causality) will be entered immediately in the appropriate AE module of the CRF. For all AEs, sufficient information will be pursued and/or obtained so as to permit i) an adequate determination of the outcome of the event (*i.e.* whether the event should be classified as a SAE); and; ii) an assessment of the casual relationship between the AE and the study treatments. Intensity of AE will be judged by the study physician, following guidelines by the European Medicines Agency (Note for Guidance on Clinical Safety Data Management).

All SAEs, unexpected adverse drug reactions or SUSARs must be reported as described in Section 6.3.

## 6.3 Reporting of serious adverse events

Any study-related unanticipated problem posing risk of harm to participants or others (including all unexpected adverse drug reactions), and any type of SAE will be immediately (within a maximum of 24 hours after becoming aware of the event) notified to the study sponsor-investigator and Co-PIs:

#### Prof. Dr. Jennifer Keiser (Sponsor-Investigator/PI)

Swiss Tropical and Public Health Institute Kreuzstrasse 2, 4123 Allschwil, Switzerland

> Tel.: +41 61 284 82 18 Fax: +41 61 284 81 05

Email: jennifer.keiser@swisstph.ch

#### Mr. Said Mohammed Ali (Co-PI)

Public Health Laboratory Ivo de Carneri P.O. Box 122 Wawi, Chake Chake, Pemba, Tanzania

Tel.: +255 24 245 20 03

E-mail: saidmali2003@yahoo.com

Within the following 48 hours, the local co-investigator must provide further information on the SAE or the unanticipated problem in the form of a written narrative to the study sponsor-investigator. This should include a copy of a completed SAE form, and any other diagnostic information that will assist the understanding of the event. In exceptional circumstances, a SAE may be reported by telephone. In these cases, a written report must be sent immediately thereafter by fax or e-mail. Names, addresses and telephone for SAE reporting will be included in the trial-specific SAE form. Relevant pages from the CRF may be provided in parallel (*e.g.*, medical history, concomitant medications).

All pregnancies in enrolled participants will be reported to the sponsor-investigator within 48 hours of becoming aware of the pregnancy. In the event of pregnancy in a treated participant, she should be monitored until the conclusion of pregnancy. The outcome of the pregnancy and any complications must be reported to the sponsor-investigator within 48 hours.

## 6.4 Safety reporting to Health Authorities, Ethics Committees and other third parties

The sponsor-investigator will send appropriate safety notifications to Health Authorities in accordance with applicable laws and regulations. Additionally, this information will be provided to the responsible ethics committee in Switzerland and Zanzibar according to national rules. Fatal or life-threatening SAEs or SUSARs will be reported within 24 hours followed by a complete report within 7 additional calendar days. Other SAEs and SUSARs that are not fatal or life-threatening will be filed as soon as possible but no later than 14 days after first knowledge by the sponsor-investigator. SAEs involving moxidectin will be reported to the manufacturer in accordance with agreements.

## 6.5 Rescue medication strategy

In case an adverse event requires medical intervention, this will be performed by the study physician and in accordance with local medical guidelines. Given the most common adverse events (headache, abdominal pain, itching, nausea, vomiting and diarrhoea), analgesics and antipyretics (*e.g.* paracetamol) are allowed to be given to participants in case of pain or fever, antiemetics (*e.g.* dimenhydrinate) to prevent nausea and vomiting and/or antibiotics to prevent or treat bacterial superinfection. In addition, electrolyte replacement solution in case of severe vomiting and diarrhoea, immunosuppressants (*e.g.* dexamethasone) in case of allergies or immune system over-reaction (*e.g.* due to a high amount of worms being expulsed) or an adsorptive antidote (*e.g.* activated charcoal) may be administered.

At the end of the study, all participants remaining positive for *T. trichiura* or any co-infection will be treated with the currently best recommended treatment.

# 7. Data management and data quality control

The investigators are responsible for an adequate data quality. Prior to the initiation of the study, a short investigator's meeting will be held between investigators of Swiss TPH and PHL-IdC. This meeting will include a detailed discussion of the protocol, performance of study procedures (standard operating procedures from previous studies available on site), CRF completion, specimen collection and diagnostic methods.

## 7.1 Source data

Source data are comprised of clinical findings and observations as well as laboratory data maintained and compiled at the study site. Source data are contained in hardcopy source documents and are allowed to be accessed by local authorities. Source data will be directly entered in the following documents:

- CRF: Primary data collection instrument for the study. It holds records of all clinical and
  physical examination data, treatment information and AEs. For every participant enrolled in the
  clinical trial a corresponding CRF exists. All data requested on the CRF must be recorded, and
  investigators will review and approve each CRF for completion.
- 2. Census: Holds name, age and sex of each potential participant.
- 3. Laboratory parasitology sheets: Record of the *T. trichiura*, *A. lumbricoides* and hookworm egg counts at all sample collection time points.
- 4. PK: Time records of PK sample collection.

## 7.2 Data collection and documentation

Data collected and produced within this trial will fall into one of the following categories:

a) Egg counts of *T. trichiura*, *A. lumbricoides* and hookworm derived from quadruplicate Kato-Katz microscopy performed at baseline as well as at 14-21 days post-treatment.

- b) Anthropometric and clinical characteristics of the trial participants collected using the study's CRF such as weight, height, blood pressure, temperature, pregnancy status (for female participants aged 10-12 years), overall health status and any abnormal medical condition or chronic disease.
- c) Finger prick blood samples for haemoglobin measurement and PK analysis.
- d) Collection date and time of each PK sample.
- e) Measured concentrations analysed from finger prick blood samples and subsequently derived PK parameters.

All data categories will be recorded paper-based (primary data source), *e.g.* on the CRF, and double-entered into the electronic data collection software REDCap (Vanderbilt University, US) using tablets. In this case, the paper-based data will represent the primary data source. All entries will be printed in blue ink and all corrections must be documented with date and initials of the respective team member. Double-entered data will be compared using the REDCap internal 'Data Comparison Tool' and any discrepancies will be reviewed against the hardcopies of the CRF and corrected accordingly. All data files in REDCap will be merged into a master file and saved as .xlsx and/or .csv file. Data analysis will be conducted with pseudonymised data and reporting of findings will be fully anonymised.

# 7.3 Ethical, legal and security issues

Information about study participants will be kept confidential and managed accordingly. Screened participants will be listed in a confidential "participant screening log" and attributed a unique participant ID (PID). In case of enrolment, participants will be listed in a confidential "participant enrolment log" utilizing the same PID. The PID will be linked with the participant's identity on a separate file (participant identification list), filed in a secured place at PHL-IdC. This document will constitute the only source to decode the pseudonymised data and will only be accessible to investigators. Personal data will be coded for data analysis. No names will be published at any time, and published reports will not allow for identification of single participants. Confidentiality will be ensured throughout the entire research project. All databases will be password secured. None of the investigators declare to have any conflicts of interest.

# 7.4 Data storage and preservation

All samples containing biological material will be destroyed after completion of the study. Paper-based and electronic source data and related material will be preserved for a minimum of 15 years to enable understanding of the study procedures, which allows the work to be assessed retrospectively and repeated if necessary. The study site (PHL-IdC) will retain the original hardcopy source documents such as CRFs to ensure that local collaborators can provide access to these documents to a monitor, auditor, or regulatory agency. Essential infrastructure such as a locked room for safe storage of hardcopy data will be made available. Electronic copies of source documents will be transferred to Swiss TPH,

Allschwil, Switzerland, for storage on secured network drives with restricted access for study personnel only. The primary storage of electronic data will be within REDCap on the Swiss TPH shared server and strictly confidential by password protection. The entire REDCap project (including all data) will be backed up regularly, *e.g.* weekly. Secondary data storage will be on personal, password-protected laptops of the PI and Co-PIs, and on a flash drive kept by Co-PIs at the study site.

# 7.5 Study documents: translations – reference language

- The protocol master document will be in English, all further language versions (*e.g.* Kiswahili) are translated thereof.
- The ICF master document will be in English, all further language versions (*e.g.* Kiswahili) are translated thereof.
- The CRF master document will be in English, all further language versions (*e.g.* Kiswahili) are translated thereof.

### 8. Statistics

## 8.1 Definition of primary endpoint

*T. trichiura* infection status 14-21 days post-treatment assessed by quadruplicate Kato-Katz is the primary endpoint in our study.

### **8.2** Justification of number of trial participants

The primary analysis of this trial aims to assess whether combined moxidectin and albendazole is more efficacious against *T. trichiura* infection compared to standard of care therapy (albendazole monotherapy) in SAC. We assumed a true CR of 30% for moxidectin-albendazole combination and 10% for albendazole monotherapy against *T. trichiura*. Assuming a loss to follow-up of 15% and requiring an allocation ratio of 3:2, we estimated that enrolling 105 participants in the moxidectin-albendazole combination arm and 70 participants in the albendazole monotherapy arm will be sufficient to identify a statistically significant difference with 85% power using a two-sided 5% significance level. Additionally, 35 individuals will be included for the placebo only arm to evaluate safety findings. In total, we anticipate to recruit 210 participants.

The suggested sample size of a maximum 5 PK samples from 24 participants (12 per moxidectin dose) is sufficiently high to determine the population PK parameters with a sparse sampling scheme.

### **8.3** Description of statistical methods

The primary analysis will use the full analysis set (available case population) according to the intention-to-treat principles defined as all randomised participants who provide any follow-up data. Only randomised participants not providing follow-up data as well as participants who were negative at

baseline and erroneously randomised will be excluded from the analysis. In addition, a per-protocol analysis will be conducted. Eligibility for analysis sets will be determined before unblinding. CRs will be calculated as the percentage of egg-positive participants at baseline who become egg-negative after treatment. Differences between CRs will be assessed by using logistic regression with only treatment and stratification variables included in the model. Results will be reported overall and by relevant stratification variable.

EPG will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the different treatment arms before and after treatment to assess the corresponding ERRs (see formula).

$$ERR = 1 - \frac{\frac{1}{n} e^{\sum \log(EPG_{follow-up} + 1)} - 1}{\frac{1}{n} e^{\sum \log(EPG_{baseline} + 1)} - 1}$$

Bootstrap resampling method with 5,000 replicates will be used to calculate 95% confidence intervals (CIs) for ERR point estimates and the difference between the ERRs.

Previous similar trials have shown that the proportion of participants lost to follow-up is usually far below 10%, therefore, no imputation of missing data will be performed. Infection status and egg counts of participants with incomplete data at follow-up (*i.e.* only one stool sample available at follow-up) will be estimated based on the available data. This means a participant is considered infected if any sample is positive and EPGs will be calculated as mean egg count of the available sample multiplied by 12.

The safety analysis set will include all treated participants. AEs will be evaluated descriptively focusing on the proportion of participants reporting symptoms before and after treatment in each arm.

Previously established nonlinear mixed-effects (NLME) models will be used to compare and determine PK parameters [21, 31]. Concentrations are measured with a validated LC-MS/MS method [31]. Using NLME, the following key PK parameters will be calculated:

- C<sub>max</sub> maximal plasma concentration
- $t_{max}$  time to reach  $C_{max}$
- AUC area under the curve, from 0 to 24 h and 0 to inf.
- $t_{1/2}$  elimination half-life

 $C_{max}$  and  $t_{max}$  will be observed values derived from the plasma concentration-time profile. Total drug exposure (AUC) and  $t_{1/2}$  will be calculated with the WinNonlin software package using compartmental analysis. The elimination half-life will be estimated by the equation:  $t_{1/2} = ln2/\lambda$ , where  $\lambda$  (the elimination rate constant) will be determined by performing a regression of the natural logarithm of the

concentration values during the elimination period. Primary PK parameters including absorption rate  $(k_a)$ , volume of distribution (V), and clearance (CL) will be estimated utilizing NLME modelling. In addition, exploratory pharmacometric PK and exposure-response analyses may be performed with the Monolix or NONMEM software package.

# 9. Duties of the investigator

# 9.1 Investigator's confirmation

This trial will be conducted in accordance with the protocol, International Conference on Harmonisation Good Clinical Practice E6 (R2) (ICH-GCP) and the current version of the Helsinki Declaration.[34, 35] All protocol modifications must be documented in writing. A protocol amendment can be initiated by either the Sponsor-Investigator/PI or any Co-PI. The Investigator will provide the reasons for the proposed amendment in writing and will discuss with the Sponsor-Investigator/PI and Co-PIs. Any protocol amendment must be approved and signed by the Sponsor-Investigator/PI and must be submitted to the appropriate Independent Ethics Committee (IEC) for information and approval, in accordance with local requirements, and to regulatory agencies if required. Approval by IEC must be received before any changes can be implemented, except for changes necessary to eliminate an immediate hazard to trial participants, or when the change involves only logistical or administrative aspects of the trial, *e.g.* change of telephone number(s).

### 9.2 Damage coverage

A general liability insurance of the Swiss TPH is in place (Winterthur Insurance, Policy No. 4746321) and a participant liability insurance has been issued in Pemba, Tanzania (National Insurance Cooperation of Tanzania LTD, Policy No. IMIS/GL/P/25/1/2024/771417).

### 9.3 Project management

The trial team will include the PI (Prof. Jennifer Keiser), three Co-PIs (Said Mohammed Ali, Viviane Sprecher, Annina Schnoz), a study physician (Dr. Ibrahim Said Mohammed), a study pharmacist (Viviane Sprecher), and a statistician (Dr. Jan Hattendorf), as well as a local medical team and several laboratory technicians. The PI and Co-PIs will be responsible for staff management, communication with the collaborative group, recruitment monitoring, data management, safety reporting, analysis, report writing and dissemination of the trial results. The Co-PIs are responsible for supervision of the lab and field technicians, staff management, participant recruitment and enrolment monitoring, supply of the material, contact to the local authorities and participating communities.

The study site (PHL-IdC) has more than 20 years of research experience with a special focus on neglected tropical diseases, including trichuriasis, and owns well-established diagnostic laboratories in parasitology and other infectious disease fields, run by trained and experienced technicians.

Infrastructure as required for the study needs will be installed as necessary before study launch. The investigator team is responsible for ensuring that the protocol is strictly followed. No changes should be made without the agreement of the PI and the Co-PIs, except when necessary to eliminate an apparent immediate hazard or danger to a study participant. All investigators will work according to the protocol and GCP. All investigators may take any steps judged necessary to protect the safety of the participants, whether specified in the protocol or not. Any such steps must be documented. During the treatment, the records are maintained by the responsible Co-PI. All entries have to be made clearly readable with a pen. All investigators must be thoroughly familiar with the properties, effects and safety of the investigational pharmaceutical product.

### 10. Ethical considerations

### **10.1** Independent Ethics Committee (IEC)

The study will be submitted for approval by the institutional research commission of Swiss TPH and the ethical committees of Switzerland and Zanzibar. The study will be undertaken in accordance with the Declaration of Helsinki and ICH-GCP.

#### 10.2 Evaluation of the risk-benefit ratio

Moxidectin and albendazole are well-known drugs and have little and mainly mild AEs as described to date (headache, abdominal pain etc.). Moxidectin is an FDA-approved drug against onchocerciasis and has been tested for trichuriasis in adolescents and adults. In the phase 1 study conducted in children and adolescents aged 4-17 years moxidectin was well tolerated in all age cohorts in the study, with no treatment-limiting adverse events identified during 24 weeks of follow-up and no adverse events leading to early study withdrawal. No adverse events were classified as serious, and no deaths were reported. Albendazole is a widely used drug in mass treatment programs against STH. All SAC enrolled in the study will benefit from a clinical examination and a treatment against STH infections. All participants remaining positive for *T. trichiura* or any co-infection will be treated with the currently best recommended treatment.

#### 10.3 Participant information and consent

All parents or caregivers of eligible participants will be asked to sign a written informed consent form. In case the parent/caregiver is illiterate, an impartial witness that can read and write has to sign the consent and the illiterate person has to give a thumb print. Parents or caregivers will have sufficient time for reflection of their child's participation. In addition, participants will be asked to sign an assent form. Information sessions in the respective communities will be conducted to explain to parents/caregivers and potential participants the purpose and procedures of the study. Informed consent forms and assent forms are orally explained in local language of the parents/caregivers and participants if necessary to ensure comprehension. Participation is voluntary and individuals have the right to withdraw from the

study at any given point in time with no further obligations. Participation itself will not be awarded with compensation.

# 10.4 Participants requiring particular protection

Our study will include SAC, since this population group is at high risk of *T. trichiura* infection. Superiority studies between moxidectin-albendazole combination and albendazole monotherapy have not been conducted to date in this population. Our trial will produce more evidence to support the search for a safe and effective treatment of trichuriasis in children and the whole community.

Throughout the entire study, from the preparation phase to the dissemination of results, community representatives (*e.g.* teachers) will be consulted to ensure any concerns regarding the study can be tackled in an anonymous and timely manner and the study addresses the community's needs as far as possible.

# 11. Quality control and quality assurance

### 11.1 Monitoring and auditing

We will work with a locally based external monitor. The monitor will conduct site visits to the investigational facilities with the purpose of monitoring the study. Details will be described in a separate monitoring plan. The investigators will grant access to study documentation, laboratory facilities, and the clinical supplies dispensing and storage area. Monitoring observations and findings will be documented and communicated to appropriate study personnel and management. A corrective and preventive action plan will be requested and documented in response to any significant deviation. No sponsor-initiated audits are foreseen, but audits and inspections may be conducted by the local regulatory authorities or ethics committees. The investigators agree to allow inspectors from regulatory agencies to review records and assist the inspectors in their duties, if requested.

### 11.2 Data and safety monitoring board (WHO) / data monitoring committee (EU/FDA)

In our study, we work with well-known drugs in a small sample size and using a single dose treatment. Nevertheless, the project advisors, Dr Said Abdallah Jongo, physician and senior clinical research scientist at the Ifakara Health Institute (IHI) in Bagamoyo, Tanzania, and Prof Dr Piero Olliaro, infectious disease physician and professor of infectious diseases associated with poverty at Oxford University, United Kingdom, will serve as independent data and safety monitoring board, they will be informed regularly and the findings discussed. This means they have the responsibility to convene, evaluate the study data and give their advice regarding the continuation or stopping of the study before the treatment, at the end of the study and in case of an important safety event.

# 12. Funding

Funding for this trial is provided by the Swiss National Science Foundation (SNSF). This funding source had no role in the design of this study and will not have any role during its execution, analyses, interpretation of the data, or decision to submit results for publication.

# 13. Dissemination of results and publication

The final results of this study will be published in a peer-reviewed scientific journal and presented at scientific conferences. SNSF will be acknowledged as study funder. All results from this investigation are considered confidential and shall not be made available to any third party by any member of the investigating team before publication. A summary of study findings may be shared with local health authorities prior to publication. After publication, study results will be made available to study participants.

# 14. References

- 1. Pullan, R.L., et al., *Global numbers of infection and disease burden of soil transmitted helminth infections in 2010.* Parasit Vectors, 2014. 7: p. 37.
- 2. World Health Organization. *Fact sheet: Soil-transmitted helminth infections*. 2023 21 August 2023]; Available from: <a href="https://www.who.int/news-room/fact-sheets/detail/soil-transmitted-helminth-infections">https://www.who.int/news-room/fact-sheets/detail/soil-transmitted-helminth-infections</a>.
- 3. US Centers for Disease Control and Prevention. *DPDx Laboratory Identification of Parasites of Public Health Concern. US Centers for Disease Control and Prevention (CDC).* 2021 [cited 2021 31 January]; Available from: <a href="https://www.cdc.gov/dpdx/index.html">https://www.cdc.gov/dpdx/index.html</a>.
- 4. Jourdan, P.M., et al., *Soil-transmitted helminth infections*. The Lancet, 2018. **391**(10117): p. 252-265.
- 5. World Health Organization, *Ending the neglect to attain the Sustainable Development Goals: a road map for neglected tropical diseases 2021–2030.* 2020, World Health Organization: Geneva.
- 6. World Health Organization, *Prevention and control of schistosomiasis and soil-transmitted helminthiasis: report of a WHO expert committee*, in *WHO Technical Report Series*. 2002, World Health Organization: Geneva.
- 7. World Health Organization, 2030 targets for soil-transmitted helminthiases control programmes. 2019, World Health Organization: Geneva.
- 8. World Health Organization, *Preventive chemotherapy in human helminthiasis Coordinated use of anthelminthic drugs in control interventions: a manual for health professionals and programme managers.* 2006, World Health Organization: Geneva.
- 9. World Health Organization, Guideline: preventive chemotherapy to control soil-transmitted helminth infections in at-risk population groups. Geneva, Switzerland. 2017, World Health Organization: Geneva.
- 10. World Health Organization, *Model List of Essential Medicines*, 22nd List. 2021, World Health Organization: Geneva.
- 11. Moser, W., C. Schindler, and J. Keiser, *Efficacy of recommended drugs against soil transmitted helminths: systematic review and network meta-analysis.* BMJ, 2017. **358**: p. j4307.
- 12. Farrell, S.H., et al., *Investigating the Effectiveness of Current and Modified World Health Organization Guidelines for the Control of Soil-Transmitted Helminth Infections*. Clin Infect Dis, 2018. **66**(suppl\_4): p. S253-S259.
- 13. Clarke, N.E., et al., Efficacy of Anthelminthic Drugs and Drug Combinations Against Soiltransmitted Helminths: A Systematic Review and Network Meta-analysis. Clin Infect Dis, 2019. **68**(1): p. 96-105.
- 14. Moser, W., C. Schindler, and J. Keiser, *Drug Combinations Against Soil-Transmitted Helminth Infections*. Adv Parasitol, 2019. **103**: p. 91-115.
- 15. Hughes, D. and D.I. Andersson, *Evolutionary consequences of drug resistance: shared principles across diverse targets and organisms.* Nat Rev Genet, 2015. **16**(8): p. 459-71.
- 16. World Health Organization, The Selection and Use of Essential Medicines Report of the WHO Expert Committee, 2017 (including the 20th WHO Model List of Essential Medicines and the 6th Model List of Essential Medicines for Children), in WHO technical report series. 2017, World Health Organization: Geneva.
- 17. Opoku, N.O., et al., Single dose moxidectin versus ivermectin for Onchocerca volvulus infection in Ghana, Liberia, and the Democratic Republic of the Congo: a randomised, controlled, double-blind phase 3 trial. The Lancet, 2018. **392**(10154): p. 1207-1216.
- 18. Keller, L., et al., *Efficacy and Safety of Ascending Dosages of Moxidectin and Moxidectin- albendazole Against Trichuris trichiura in Adolescents: A Randomized Controlled Trial.* Clin Infect Dis, 2020. **70**(6): p. 1193-1201.
- 19. Welsche, S., et al., Efficacy and safety of moxidectin and albendazole compared with ivermectin and albendazole coadministration in adolescents infected with Trichuris trichiura in Tanzania: an open-label, non-inferiority, randomised, controlled, phase 2/3 trial. Lancet Infect Dis, 2023. 23(3): p. 331-340.

- 20. Sprecher, V.P., et al., Efficacy and Safety of Moxidectin-Albendazole and Ivermectin-Albendazole Combination Therapy Compared to Albendazole Monotherapy in Adolescents and Adults Infected with Trichuris trichiura: A Randomized, Controlled Superiority Trial. Clin Infect Dis, 2023. 77(9): p. 1294-1302.
- 21. Opoku, N.O., et al., Safety and pharmacokinetics of a single oral dose of moxidectin in subjects aged 4 to 17 years with (or at risk of) onchocerciasis, to identify an optimal dose for treatment of children 4 to 11 years: Results of an open label study. ASTMH 2022 Annual Meeting Abstract Book, 2022: p. 12.
- 22. Geary, T.G., et al., *Unresolved issues in anthelmintic pharmacology for helminthiases of humans*. Int J Parasitol, 2010. **40**(1): p. 1-13.
- 23. Oshikoya, K.A., H.M. Sammons, and I. Choonara, *A systematic review of pharmacokinetics studies in children with protein-energy malnutrition*. European Journal of Clinical Pharmacology, 2010. **66**(10): p. 1025-1035.
- 24. Katz, N., A. Chaves, and J. Pellegrino, *A simple device for quantitative stool thick-smear technique in schistosomiasis mansoni*. Rev Inst Med Trop São Paulo, 1972. **14**(6): p. 397-400.
- 25. Dacombe, R.J., et al., *Time delays between patient and laboratory selectively affect accuracy of helminth diagnosis.* Trans R Soc Trop Med Hyg, 2007. **101**(2): p. 140-5.
- 26. Nikolay, B., S.J. Brooker, and R.L. Pullan, Sensitivity of diagnostic tests for human soil-transmitted helminth infections: a meta-analysis in the absence of a true gold standard. Int J Parasitol, 2014. **44**(11): p. 765-74.
- 27. Martin, L.K. and P.C. Beaver, *Evaluation of Kato Thick-Smear Technique for Quantitative Diagnosis of Helminth Infections* \*. The American Journal of Tropical Medicine and Hygiene, 1968. **17**(3): p. 382-391.
- 28. Bergquist, R., M.V. Johansen, and J. Utzinger, *Diagnostic dilemmas in helminthology: what tools to use and when?* Trends Parasitol, 2009. **25**(4): p. 151-6.
- 29. Presland, S.L., E.R. Morgan, and G.C. Coles, *Counting nematode eggs in equine faecal samples*. Vet Rec, 2005. **156**(7): p. 208-10.
- 30. Cooke, I.R., et al., *Analysis of menisci formed on cones for single field of view parasite egg microscopy*. J Microsc, 2015. **257**(2): p. 133-41.
- 31. Hofmann, D., S. Sayasone, and J. Keiser, *Development and validation of an LC-MS/MS method* for the quantification of the anthelmintic drug moxidectin in a volumetric absorptive microsample, blood, and plasma: Application to a pharmacokinetic study of adults infected with Strongyloides stercoralis in Laos. J Chromatogr B Analyt Technol Biomed Life Sci, 2021. **1166**: p. 122556.
- 32. World Health Organization, *Haemoglobin concentrations for the diagnosis of anaemia and assessment of severity (WHO/NMH/NHD/MNM/11.1)*. 2011, Vitamin and Mineral Nutrition Information System: Geneva.
- 33. International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use: ICH Harmonised Tripartite Guideline. Clinical Safety Data Management: definition and standards for expedited reporting E2A. 1994.
- 34. International Council for Harmonization (ICH), *Integrated addendum to ICH E6(R1): Guideline for good clinical practice E6(R2)*. 2016, International council for harmonisation of technical requirements for pharmaceuticals for human use (ICH): Geneva, Switzerland.
- 35. World Medical Association (WMA), WMA Declaration of Helsinki Ethical principles for medical research involving human subjects. 2013, World Medical Association: Fortaleza, Brazil.